CLINICAL TRIAL: NCT02854267
Title: Organ Procurement : Usefulness of a Guide for Meeting With the Next of Kin
Acronym: CANEVAS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CANEVAS
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Organ Donation
Keywords: organ procurement; brain death; organ donation; next of kins
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group without guide, before guide's diffusion: For this group, only the primary endpoint (refusal rate) will be assessed, using the French Biomedicine Agency database; The group without guide is made up by all registered situations of brain death patients on the database (nationwide) minus the situations occuring in the group with guide (22 intensive care units forming the 'RESEAU NORD FRANCILIEN' network). The period before the diffusion of the guide is from 1st of july 2012 to 30th of june 2014
- group without guide, after guide's diffusion: For this group, only the primary objective (refusal rate) will be assessed, using the French Biomedicine Agency database; The group without guide is made up by all the registered situations of brain death patients on the database minus the situations occuring in the group with guide ('RESEAU NORD FRANCILIEN'). The period after the diffusion of the guide is from 1st of january 2017 to 31st of december 2018
- Group with guide, before guide's diffusion: For this group, only the primary endpoint (refusal rate) will be assessed, using the French Biomedicine Agency database; The group with guide is made up by all the registered situations of brain death patients on the database occuring in the 22 intensive care unit forming the 'RESEAU NORD FRANCILIEN' network. The period after the diffusion of the guide is from 1st of january 2017 to 31st of december 2018.
- Group with guide, after guide's diffusion: For this group, the primary endpoint (refusal rate) will be assessed, using the French Biomedicine Agency database. The secondary endpoints (level of anxiety of the caregivers before the meeting with the next of kins as measured by the french short version of Spielberger test and compliance to the guide) will be assessed by the datasheet prospectively filled by the caregivers. The group with guide is made up by all the registered situations of brain death patients on the database occuring in the 22 intensive care unit forming the 'RESEAU NORD FRANCILIEN' network. The period after the diffusion of the guide is from 1st of january 2017 to 31st of december 2018

SUMMARY:
A dedicated guide for physicians and organ procurement nurses meeting with the next of kin could be associated with a reduction in organ donation refusal rate, and in anxiety of professionals involved in such meetings

DETAILED DESCRIPTION:
The main obstacle for organ procurement in brain dead patients in France is organ donation refusal by the next of kin. When refusal is reflecting the patient's position, ending the organ donation procedure respects the bioethic French laws. Nevertheless, the actual position of the deceased patient often remains unknown. In these cases, organ donation refusal does not necessarily respect the deceased wishes. Many factors have been associated to next of kin organ donation refusal in such situations. Among those factors, some concerning the meeting with the next of kin have been isolated. French data on this subject are lacking.

A dedicated guide for the conduct of meetings with the next of kin has been elaborated by a working group of our network. Its diffusion will take place last quarter of 2016. The purpose of our study is to evaluate its usefulness through an observational multicenter before-after study, concerning every situation of brain dead patient where the next of kin are met by the medical staff. The refusal rate will be assessed over the first period (before the diffusion of the guide), from july 2012 to june 2014, and compared to that assessed over the second period (after the diffusion of the guide) from january 2017 to december 2018, using the national database of Biomedicine Agency. A comparison of this change in refusal rate will be made between centers of our network and the remaining centers in France nationwide. Anxiety of professionals will be assessed prospectively after each meeting conducted in one of our network centers, over 2 periods, before (from July to October 2016) and after (starting in january 2017) the diffusion of the dedicated guide for the conduct of the meeting with the next of kin. Compliance to the guide by the physicians and organ procurement nurses will be assessed after its diffusion in the centers of our network.

ELIGIBILITY:
Inclusion Criteria:

* situation of confirmed brain dead patient, or dead patient with pending confirmation of brain death

Exclusion Criteria:

* situations where the next of kins are met before brain death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Interviews with next of kins as a part of organ donation
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Refusal to organ procurement as expressed by next of kins | 2 years
  Assessed in the national biomedicine agency database retrospectively over a 2-years period before diffusion of a dedicated guide for meeting, and prospectively over a 2 years period after the diffusion of a dedicated guide for meeting

SECONDARY OUTCOMES:
Anxiety level of caregivers after meeting with the next of kins | 2 years
  The anxiety will be measured by the short French version of the Spielberger anxiety state scale, and assessed prospectively over 2 periods, before and after the diffusion of a dedicated guide for meeting
Compliance to the guide | 2 years
  The compliance will be measured though a debriefing form filled by the caregivers after each meeting with the next of kins

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Kandelman, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided